CLINICAL TRIAL: NCT01389050
Title: Use of High Precision Radiotherapy in the Management of Soft-Tissue Sarcomas
Brief Title: High Precision RT For Soft-Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 10-0854-CE
Record Dates: First submitted 2011-06-30; First posted 2011-07-07 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Soft-Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up (No Intervention): Data from these patients will be added to retrospectively gathered data from the PMH radiotherapy data bank (approximately 50 patients). The data collected will be analyzed using descriptive statistics.
- Prospective (Experimental)
  Interventions: Radiation: Intensity-Modulated Radiotherapy; Radiation: Daily Cone Beam CT

INTERVENTIONS:
Radiation: Intensity-Modulated Radiotherapy — Radiotherapy for the treatment of retroperitoneal sarcoma. IMRT will be 50.4 Gy given in 28 fractions.
  Other Names: Pre-operative IMRT
  Arms: Prospective
Radiation: Daily Cone Beam CT — Images and information from the daily CT will be used for the repositioning of the patient prior to their treatments as per standard procedures.
  Other Names: daily cone-beam Computed Tomography (CT)
  Arms: Prospective

SUMMARY:
This research study aims at defining 1) how retroperitoneal sarcomas change over the course of radiotherapy and 2) how radiotherapy affects your well-being. While the investigators know that radiotherapy before surgery is safe and effective, the amount of tumor motion and size change during radiotherapy is unknown. There is also very little information that describes the side-effects of radiotherapy in the treatment of this disease.

DETAILED DESCRIPTION:
Soft-tissue sarcomas (STS) that arise from the retroperitoneum are rare malignancies that are anatomical located deep within the abdominal area and thus pose challenges to surgical and radiotherapeutic management of the patient. As a result, the local control and overall survival for patients with retroperitoneal sarcomas (RPS) are worse than STS from the extremities. Current treatment strategy involves pre-operative radiotherapy followed by surgery. Use of intensity-modulated radiotherapy (IMRT) in RPS had allowed for more conformal treatments with the aim of sparing normal tissues from high doses of irradiation. Yet the accuracy and coverage of IMRT depend highly on target motion, and little is known about the motion of RPS during the course of radiotherapy. As well, RPS are commonly in close proximity to sensitive organs for which the long-term toxicity and effect on quality of life secondary to radiation is unknown. The current study seeks to evaluate the extent of tumor motion during radiotherapy and the impact of radiotherapy to patient toxicity and quality of life. At the conclusion of this study, our results will hopefully identify the optimum PTV, the importance of different normal tissues and their dose-volume constraints, the role of image guidance, and the potential for dose escalation in the treatment of RPS.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of sarcoma (except for GIST, Ewing's sarcoma and rhabdomyosarcoma) within the retroperitoneum. These include patients with locally recurrent disease
* Planned to receive pre-operative radiotherapy
* Will undergo a planning CT
* Karnofsky Performance Status of ≥ 70 within 28 days prior to study entry
* No systemic chemotherapy given prior to pre-operative radiotherapy
* Able to provide written, informed consent
* Women of childbearing potential and men who are sexually active must practice adequate contraception.

Exclusion Criteria:

* Tumor pathology of GIST, Ewing's sarcoma or rhabdomyosarcoma
* Metastatic disease to the retroperitoneum from a primary sarcoma not originating from the retroperitoneum
* Systemic chemotherapy given prior to pre-operative radiotherapy.
* Intent on giving chemotherapy ≤ 12 months from the completion of radiotherapy
* Inability to undergo a 4D-CT simulation
* KPS < 70
* Unable to provide informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
To determine the extent of inter-fractional and intra-fractional movement of the GTV during radiotherapy treatments. | 3 years
  To quantify and describe the movement of the tumor during and between radiotherapy treatments using imagings acquired during the course of radiotherapy planning and treatments.
To assess the acute and long-term toxicity of pre-operative radiotherapy as a function of the dose given to normal tissues and its impact on patient quality of life. | 10 years
  To describe the effect of radiotherapy to the patient by measuring the acute and long-term side-effects of radiation therapy.

SECONDARY OUTCOMES:
Describe variations in the volume and shape of the GTV over the course of the treatment and need for adaptive therapy. | 3 years
  To measure and better define the response of the tumor to radiotherapy during treatments.
Correlate the pattern of local recurrence with the dose of radiation delivered accounting for motions and volume changes of target structures. | 10 years
  To determine whether there is a pattern of local relapse with the actual dose of radiation delivered to the tumor environment when tumor volumetric and positional changes are taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Catton, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada